CLINICAL TRIAL: NCT05077293
Title: BETTER CARE-HF Pilot Study: Building Electronic Tools To Enhance and Reinforce CArdiovascular REcommendations - Heart Failure, a Pilot Study
Brief Title: Building Electronic Tools To Enhance and Reinforce Cardiovascular Recommendations - Heart Failure
Acronym: BETTER CARE-HF
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: QI-BETTER CARE-HF PS
Record Dates: First submitted 2021-10-03; First posted 2021-10-14 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: Best Practice Alert; In-Basket message; Mineralocorticoid Receptor Antagonists; MRA; guideline-directed medical therapy; GDMT
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Best Practice Alert group: Providers will receive a BPA at the time of visit for patients with HFrEF who are not on MRA (and who do not have contraindication to MRA). This alert will be visible on the first screen displayed in the electronic health record and will display the patient's current HFrEF therapies, EF, blood pressure, potassium, and glomerular filtration rate. The alert will give access to an outpatient heart failure order set, and also provide links to the most recent guidelines.
  Interventions: Other: Best Practice Alert (BPA)
- In-Basket Message group: Providers will receive a biweekly in-basket messages linking to a list of patients who have been seen in the past year with HFrEF who are not on MRA (and who do not have contraindication to MRA). This list will display each patient's current hFrEF therapies, EF, blood pressure, potassium, glomerular filtration rate, and date of last visit. From the list, providers can access the patient's chart, order medications, and document communication with the patient.
  Interventions: Other: In-Basket Message
- Control group: Patients who will receive the current standard practice of care (no alerts)

INTERVENTIONS:
Other: Best Practice Alert (BPA) — A BPA will fire in the EHR reminding care providers of the best practice when prescribing medical therapies for heart failure patients.
  Groups: Best Practice Alert group
Other: In-Basket Message — An In-Basket message will be sent biweekly to care providers with a reminder of the best practice when prescribing medical therapies for heart failure
  Groups: In-Basket Message group

SUMMARY:
This is a feasibility study using a cross-over design to implement and compare a best practice alert (BPA) with an automated in-basket message to inform providers when a patient with heart failure and reduced ejection fraction (HFrEF) is not on appropriate medical therapy. The data from this pilot study will lead to a randomized controlled trial to compare the effectiveness of the BPA versus an automated in-basket message, versus usual care (no intervention).

DETAILED DESCRIPTION:
An estimated 68,000 deaths per year nationwide can be attributed to gaps in care for patients with heart failure and reduced ejection fraction (HFrEF), with the majority being due to lack of mineralocorticoid receptor antagonists (MRA). Despite proven benefits in randomized trials, class I guideline recommendations, and published clinical performance measures, patients with HFrEF are often not on guideline-directed medical therapy (GDMT). While successful interventions for improvement in prescription of GDMT have often included multidisciplinary approaches with dedicated staff, the relatively high cost of hiring additional personnel has led to an interest in electronic health record (EHR)-based interventions. Prior studies on EHR-based interventions in this arena have mainly been conducted in the inpatient setting, which is limited to one encounter during acute hospitalization, a setting often complicated by renal dysfunction or hypotension that can limit prescription of MRA. The development and study of outpatient EHR-based alerts for HFrEF GDMT are needed. Two types of outpatient EHR-based interventions include best practice alerts (BPA) and automated in-basket messages. Both of these methods have limited data, with some studies showing benefit and others demonstrating provider fatigue and burnout. To our knowledge, there is no study that has directly compared these different types of EHR-based interventions.

This is a feasibility study using cross-over design at two outpatient clinics in a large health system to implement and compare a best practice alert (BPA) and an automated in-basket message to inform providers when a patient with heart failure and reduced ejection fraction (HFrEF) is not on appropriate medical therapy. The data from this study will lead to a randomized controlled trial to compare the effectiveness of the BPA versus an automated in-basket message, versus usual care (no intervention).

ELIGIBILITY:
Inclusion Criteria:

* Cardiologist visit
* Transthoracic echocardiogram with the most recent EF >= 40%

Exclusion Criteria:

* Hypotension: SBP < 95
* Hyperkalemia: most recent K > 5.1, or any K >5.5
* Renal dysfunction: eGFR < 30
* Ventricular assist device
* Hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Langone cardiology outpatients
Sampling Method: Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients prescribed MRA | 14 days after alert
Incidence of provider engagement with each alert type | 14 days after alert
  Provider engagement is reported when the provider clicks on links or buttons within each alert.

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone Health, New York, New York, United States